CLINICAL TRIAL: NCT02950415
Title: Does Virtual Parental Presence Reduce Preoperative Anxiety in Children: A Randomized Controlled Trial
Brief Title: Does Virtual Parental Presence Reduce Preoperative Anxiety in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Clyde Matava, Staff Anesthesiologist, The Hospital for Sick Children
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: 1000053821
Record Dates: First submitted 2016-08-30; First posted 2016-11-01 (Estimated); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Restraint, Physical

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- virtual + coaching (Other): Parent is present virtually via an internet pad (iPad) and has received coaching about how best to verbally soothe child
  Interventions: Behavioral: virtual; Behavioral: coaching
- virtual + no coaching (Other): Parent is present virtually via an internet pad (iPad) and has not received coaching about how best to verbally soothe child
  Interventions: Behavioral: virtual; Behavioral: no coaching
- physical + coaching (Other): Parent is physically present and has received coaching about how best to verbally soothe child
  Interventions: Behavioral: coaching; Behavioral: physical
- physical + no coaching (Other): Parent is physically present and has not received coaching about how best to verbally soothe child
  Interventions: Behavioral: physical; Behavioral: no coaching

INTERVENTIONS:
Behavioral: virtual — Parent is present via an internet pad (iPad)
  Arms: virtual + coaching; virtual + no coaching
Behavioral: coaching — Parent learns what to say verbally to soothe child
  Arms: physical + coaching; virtual + coaching
Behavioral: physical — Parent is present in the operating room
  Arms: physical + coaching; physical + no coaching
Behavioral: no coaching — Parent does not learn what to say verbally to soothe child
  Arms: physical + no coaching; virtual + no coaching

SUMMARY:
Children undergoing anesthesia are often very frightened by the experience. This can lead to bed wetting, nightmares and stranger anxiety that can last for weeks. Moreover, this can influence their future experiences with anesthesia and surgery. The investigators believe the presence of a parent via video might work better as parental fear is not transferred to the child. The investigators also believe that parents who are coached on how to assist their child during anesthesia will have a better impact. As such the investigators are carrying out this study to assess whether parents who are coached and are present in either video or physical form will be more effective in reducing anxiety at induction of anesthesia.

DETAILED DESCRIPTION:
The investigators' goal in this study is to investigate the effects of virtual parental presence and coaching of parents on anxiety in children at induction of anesthesia. The primary hypothesis is virtual parental presence during induction of anesthesia is superior to physical parental presence during induction of anesthesia in reducing anxiety in children at induction of anesthesia. The secondary hypothesis is that the coaching of parents modulates the effect of physical or video parental presence at induction anesthesia on children's anxiety.

ELIGIBILITY:
Inclusion Criteria:

1. Children from ages 18 months to 12 years old
2. American Society of Anesthesiologists physical status I, II or III
3. No previous exposure to anesthesia or surgery
4. Same Day surgery
5. English speaking parents and child

Exclusion Criteria:

1. Children with developmental delay
2. Children with psychological / emotional disorders
3. Children with language barrier
4. Previous anesthetic or surgical experience
5. Children whose eyes will be closed following surgery
6. Children on sedative or psychoactive medication
7. History of allergy to medications in our study
8. Children with expected difficult intubation
9. Children presenting for emergency surgery
10. Family history or personal history of malignant hyperthermia / risk of malignant hyperthermia
11. Consent not obtained or withdrawal of consent
12. Children who are violent during induction of anesthesia
13. Cancellation of surgery

Ages: 18 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2017-05-16 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Anxiety in children | Day of surgery, immediately following consent
  measured using the modified Yale Preoperative Anxiety Scale (mYPAS)
Change in child anxiety | Day of surgery, immediately preceding surgery
  measured using the modified Yale Preoperative Anxiety Scale (mYPAS)

SECONDARY OUTCOMES:
Induction compliance | Day of surgery, immediately preceding surgery
  measured using the Induction Compliance Checklist
Child temperament | Day of surgery, immediately following consent
  measured using the Emotionality Activity Sociability Impulsivity Instrument of Child Temperament (EASI)
Parental anxiety | Day of surgery, immediately following consent
  measured using the State-Trait Anxiety Inventory (STAI)
Change in parental anxiety | Day of surgery, immediately preceding surgery
  measured using the State-Trait Anxiety Inventory (STAI)
Parental satisfaction | Day of surgery, five minutes after surgery has commenced
  measured using The Hospital for Sick Children satisfaction questionnaire
Anesthesiologist satisfaction with task load | Day of surgery, immediately following surgery
  measured using the NASA Task Load Index (NASA-TLX)
Anesthesiologist satisfaction with technology usability | Day of surgery, immediately following surgery
  measured using the System Usability Scale (SUS)
Induction nurse satisfaction with task load | Day of surgery, immediately following surgery
  measured using the NASA Task Load Index (NASA-TLX)
Induction nurse satisfaction with technology usability | Day of surgery, immediately following surgery
  measured using the System Usability Scale (SUS)
Anesthetic requirements | Day of surgery, intra-operatively
  measurement includes recording dose of anesthetic(s) used
Anesthetic requirements | Day of surgery, from time of randomisation up to 4 hours afterwards
  includes recording dose of anesthetic(s) used on a data collection form
Post-hospitalization negative behaviours | Two to three days after surgery
  measured using the Posthospitalization Behaviour Questionnaire (PHBQ)

CONTACTS AND LOCATIONS:
Overall Officials: Clyde Matava, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No